CLINICAL TRIAL: NCT05109377
Title: Endocan Level in Patients With Erectile Dysfunction and Relationship With Tadalafil Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Veysel Bayburtluoğlu, Principal Investigator, Ankara Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: E-93471371-514.10
Record Dates: First submitted 2021-09-04; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Erectile Dysfunction
Keywords: Endocan; Erectile dysfunction; Tadalafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5mg tadalafil (Other): 5mg tadalafil
  Interventions: Diagnostic Test: Endocan; Drug: tadalafil
- 20mg tadalafil (Other): 20 mg tadalafil
  Interventions: Diagnostic Test: Endocan; Drug: tadalafil

INTERVENTIONS:
Diagnostic Test: Endocan — Endocan will measured before and after treatment
Drug: tadalafil — tadalafil

SUMMARY:
The investigators analyze the patients' endocan levels, IIEF scores, and hormon levels both before and after tadalafil (5 or 20mg) treatment. The investigators want to see erectile dysfunction severity and tadalafil treatment relations with endocen level.

DETAILED DESCRIPTION:
The investigators will include at least 90 patients in study. Blood tests will taken before and after tadalafil treatment and will store at -80 celcius degree.

ELIGIBILITY:
Inclusion Criteria:

• Patients with erectile dysfuction

Exclusion Criteria:

* Psychogenic erectile dysfunction
* Erectile dysfunction associated with hormonal disorders
* Drug related erectile dysfunction

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2021-11-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Rates of IIEF Score | 1 month
  Levels of Endocan relationship with IIEF

SECONDARY OUTCOMES:
Levels of Endocan | 1 month
  Levels of Endocan with tadalafil treatment

CONTACTS AND LOCATIONS:
Overall Officials: Veysel Bayburtluoğlu, Principal Investigator — Ministry of Health
Locations (1):
- Veysel Bayburtluoğlu, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Research data